CLINICAL TRIAL: NCT03553511
Title: Short and Long-term Outcomes After Total Laparoscopic Hysterectomy With Vaginal Vault Suspension to the Uterosacral Ligaments Versus Vaginal Hysterectomy With McCall Culdoplasty for the Treatment of Stage II-III Pelvic Organ Prolapse.
Brief Title: Laparoscopic Hysterectomy With Vaginal Vault Suspension to the Uterosacral Ligaments for Stage II-III Pelvic Organ Prolapse.
Acronym: LULS-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Medical Doctor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LULS-1
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: Laparoscopy; Hysterectomy; Uterosacral ligaments suspension; McCall culdoplasty; Post-hysterectomy vault prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uterosacral ligaments suspension (Experimental): Women affected by stage II-III pelvic organ prolapse undergoing total laparoscopic hysterectomy with vaginal vault suspension to the uterosacral ligaments.
  Interventions: Procedure: Vaginal vault suspension to the uterosacral ligaments
- McCall culdoplasty (Active Comparator): Women affected by stage II-III pelvic organ prolapse undergoing vaginal hysterectomy with McCall culdoplasty.
  Interventions: Procedure: McCall culdoplasty

INTERVENTIONS:
Procedure: Vaginal vault suspension to the uterosacral ligaments — Laparoscopic hysterectomy with vaginal vault suspension to the uterosacral ligaments
  Arms: Uterosacral ligaments suspension
Procedure: McCall culdoplasty — Vaginal hysterectomy with McCall culdoplasty
  Arms: McCall culdoplasty

SUMMARY:
The International Continence Society defines post-hysterectomy vault prolapse (PHVP) as descent of the vaginal cuff scar below a point that is 2 cm less than the total vaginal length above the plane of the hymen. The incidence of PHVP has been reported to affect up to 43% of hysterectomies. The risk of prolapse following hysterectomy is 5.5 times more common in women whose initial hysterectomy was for pelvic organ prolapse as opposed to other reasons.

Techniques available to manage PHVP aim to ultimately suspend the vaginal vault. Approaches include vaginal, e.g. uterosacral ligament suspension, sacrospinous ligament fixation, open procedures and more recently laparoscopic, e.g. sacrocolpopexy and uterosacral plication.

Data published so far do not allow to draw a firm conclusion about the best treatment to prevent PHVP for women undergoing hysterectomy for stage II-III pelvic organ prolapse. Considering this scenario, in the current study the investigators aim to evaluate short and long-term outcomes after total laparoscopic hysterectomy with vaginal vault suspension to the uterosacral ligaments versus vaginal hysterectomy with McCall culdoplasty for the treatment of stage II-III pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-III pelvic organ prolapse
* Bilateral preservation of the ovaries
* Sexually active women

Exclusion Criteria:

* Smoking
* Body Mass Index > 30
* Strenuous activity (frequent heavy lifting)
* Other gynecological and non-gynecological (chronic endocrine, metabolic, autoimmune, neoplastic diseases) comorbidities
* Pharmacological and/or nonpharmacological treatment (including pelvic floor exercises) in the six months preceding the surgery or during the study period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 12 months after surgery
  Vaginal vault prolapse

SECONDARY OUTCOMES:
Urinary impact questionnaire score (total score minimum: 0, maximum: 100) | 12 months after surgery
  A specific questionnaire developed to investigate the impact of urinary symptoms and signs on the quality of life.
Pelvic Organ Prolapse Impact Questionnaire (total score minimum: 0, maximum: 100) | 12 months after surgery
  A specific questionnaire developed to investigate the impact of prolapse-related symptoms and signs on the quality of life.
Colorectal-Anal Impact questionnaire (total score minimum: 0, maximum: 100) | 12 months after surgery
  A specific questionnaire developed to investigate the impact of prolapse-related colorectal and anal symptoms and signs on the quality of life.
Prolapse/urinary incontinence sexual questionnaire score (total score minimum: 0, maximum: 48) | 12 months after surgery
  A specific questionnaire developed to investigate the impact of prolapse/urinary incontinence on sexual functions.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria; Jvan Casarin, M.D., Principal Investigator — Università degli Studi dell'Insubria; Antonella Cromi, M.D., Ph.D., Study Chair — Università degli Studi dell'Insubria; Fabio Ghezzi, M.D., Study Director — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided